CLINICAL TRIAL: NCT06545123
Title: Unraveling the Impact of Distinct Exercise Modalities on GUT Microbiome and Gut-derived Metabolites in Older Adults with Sarcopenia
Brief Title: Distinct Exercise Modalities on Gut Microbiome
Acronym: DEMGUTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faculty of Sports- Research Center in Physical Activity, Health and Leisure (Other)
Collaborators: Unit for Multidisciplinary Research in Biomedicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEFADE 04 2024
Record Dates: First submitted 2024-07-20; First posted 2024-08-09 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Sarcopenia; Older Adults
Keywords: Gut Microbiome; Exercise; Metabolomics; Physical function
MeSH Terms: conditions — Sarcopenia; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants that meet the inclusion/exclusion criteria will be randomly assigned to: i) moderate aerobic exercise (AER); ii) resistance exercise (RES); or iii) concurrent exercise training (RES+AER).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Resistance exercise training (Active Comparator): The main part of RES group session will include free weights, weight machines and calisthenics. Loads will be set and adjusted based on 1 repetition maximum (1RM) method (details are described in Table 2). Exercises will be standardized but exercises may be adapted according to participants limitations. For RES group, the intervention was divided in 2 periods: a) 3- weeks adaptation phase (7-10 exercises; 1-2 sets; 15-20 reps; 40-60% 1RM); b) 9-weeks training phase (8 exercises; 3 sets; 6-12 reps; 70% 1RM; intensity measured by the rate of perceived exertion (RPE) 3-5 on category ratio 10 (CR10) scale progressing to RPE 6-8; resting 60-120 s between sets; 3-5 min between exercises) as recommended (29). Each session will aim at two anatomical regions (upper limbs, torso, back, lower limbs).
  Interventions: Behavioral: Concurrent exercise training
- Aerobic exercise training (Active Comparator): The main part of AER group sessions will include treadmill, stationary and elliptical bikes. The intensity throughout these sessions will be measured by heart rate maximum (HRmax) and by RPE 3-5 on CR10 scale progressing to RPE 6-8. The main part of AER group was divided in 3 periods; a) from week 1-2 (50% HRmax: 3x15 min+3min rest); b) week 3-4 (60% HRmax: 2x23min+5min rest); c) week > 5 (70% HRmax: continuous).
  Interventions: Behavioral: Concurrent exercise training
- Concurrent exercise training (Active Comparator): The main part of RES+AER group sessions will combine both exercise training protocols. The main parts of this group will start with resistance training using weights, weight machines and calisthenics combined with a main part of moderate aerobic exercises in the treadmill, stationary and elliptical bikes. This intervention was divided into 2 phases: a) a 3-week adaptation period (4-6 exercises; 1-2 sets; 15-20 reps; 40-60% 1RM); b) 9-weeks training phase (4 exercises; 3 sets; 6-12 reps; 60-70% 1RM; intensity measured by the RPE 3-5 on CR10 scale progressing to RPE 6-8; resting 60-120 s between sets; 3-5 min between exercises). Afterward, the moderate aerobic exercise training part will include three phases: 50% HRmax: 1x15 min); b) week 3-4 (60% HRmax: 1x23min); c) week > 5 (70% HRmax: continuous).
  Interventions: Behavioral: Concurrent exercise training

INTERVENTIONS:
Behavioral: Concurrent exercise training — The experimental groups (AER, RES and AER+RES) will be enrolled in a supervised center-based exercise program for 12 weeks (3 days/week; 60 min/d). Sessions will occur in the morning, on alternating days of the week, and will be supervised by experienced exercise physiologists

SUMMARY:
Sarcopenia is a multifactorial muscular disease with detrimental clinical consequences, impairing physical function, functional independence, quality of life, need for long-term care and premature mortality. The development of sarcopenia is influenced by a complex interaction of multiple environmental and endogenous factors. However, to date, these complex mechanisms were unable to fully explain sarcopenia adverse health outcomes on skeletal muscle mass and function in older adults. Recently, the gut microbiome and its gut-derived metabolites have emerged as a key player in sarcopenia, with evidence suggesting that influence many underlying pathophysiological mechanisms (i.e., immune and inflammation system, anabolic resistance, insulin sensitivity, and energy production) that are involved in the development of sarcopenia. Current treatment guidelines of sarcopenia reinforce the role of exercise training, particularly resistance training to prevent adverse health outcomes. Exercise also stimulates favorable changes in gut microbiome composition and function, leading to host health benefits, regardless of nutrition. Nonetheless, the effects of exercise training on gut microbiome in patients with sarcopenia remains unclear, with existing evidence derived mainly from observational studies. In addition, the available evidence suggests that different types of exercise modalities may elicit distinct changes in gut microbiota composition but, to date, no study specifically addressed the optimal type of exercise modality in older adults considering the impact of gut microbiota composition or of gut-derived metabolites. Thus, despite the growing body of literature on the gut-muscle axis and sarcopenia, evidence from comparative studies focused on different exercise training regimens with a randomized controlled trial design in the impact of gut microbiota on skeletal muscle mass and function in sarcopenic patients is still lacking. Given that aerobic and resistance exercise stimulate different bioenergetic mechanisms and metabolic signaling pathways, we hypothesize that gut microbiome composition may be differently modulated by these distinct exercise regimens and that differently impact skeletal muscle mass and function, and physical performance in older adults. Leveraging current recruitment, logistics and human resources from a community exercise training program and the internal institutional collaborations, the investigative team will build a consecutive line of research to fill this literature gap and explore the impact of different exercise regimens on gut microbiome composition and gut-derived metabolites in these patients. The research team will start with a pilot single center 3-parallel arm open-label randomize control trial. Participants that meet the inclusion/exclusion criteria will be randomly assigned to: i) moderate aerobic exercise (AER); ii) resistance exercise (RES); or iii) concurrent exercise training (RES+AER). Participants in the experimental groups will engage in a supervised center-based exercise intervention (12-weeks, 3d/w, 60min/d). All participants will be assessed at i) baseline, ii) end of intervention (14 weeks) and iii) at close-out (26-weeks). The primary outcome will be the change in the relative abundance of Faecalibacterium prausnitzii and other SCFA producing bacteria after the intervention (14-weeks). Secondary outcomes include 1) change of Faecalibacterium prausnitzii relative abundance at close-out (26 weeks); 2) change of relative abundance of Lactobacillus and Bifidobacterium genera after the intervention and at the end of the follow-up. A set of complementary outcomes will also be assessed to broadly characterize the impact of each exercise intervention, including body composition, skeletal muscle function, functional performance and general gut microbiome composition. Other important confounding outcomes will be evaluated, including nutritional intake, daily physical activity, medication and supplementation use, and associated comorbidities. In the long term, the study team expects to contribute to clinical guidance and exercise prescription in older adults with sarcopenia using an evidence-based approach by exploring the optimal exercise mode to elicit favorable gut and skeletal muscle health benefits.

DETAILED DESCRIPTION:
The gut microbiome is an important regulator of metabolism and has recently emerged as a relevant contributor to musculoskeletal health and disease, specifically to changes in skeletal muscle mass and function through a communication axis known as the gut-muscle axis. This posited gut-muscle communication pathway raises the attractive possibility that by manipulating the gut microbiota composition and function, scientists could mediate changes in skeletal muscle health and prevent sarcopenia adverse health outcomes. Thus, therapeutic strategies developed to modulate gut microbiome composition may have clinically meaningful implications in age-related muscle loss and physical function decline. Exercise has been shown to modulate the gut microbiome in older adults, but the evidence from well-designed randomized clinical trials is scarce. On the one hand, current guidelines recommend resistance training to reduce age-related skeletal muscle loss and physical function impairment. Still, on the other hand, aerobic exercise training is associated with increased microbiota diversity and an increase in SCFA-producing taxa, which has been linked to skeletal muscle health benefits and improved function. Given that these two exercise training regimens have different bioenergetic pathways, the study team hypothesized that each regimen promotes distinct alterations in gut microbiome composition. In contrast, combining both forms of exercise (resistance + aerobic) may lead to an added effect. Therefore, unraveling the impact of these exercise regimens on the gut microbiome is crucial to fill this relevant knowledge gap and to help clarify the optimal exercise regimen to manage sarcopenia. The research team long-term goal is to develop a consecutive line of research to explore the impact of these different exercise training regimens (i.e., resistance, aerobic, and concurrent exercise training) on gut microbiome composition and gut-derived metabolites and investigate its effects on skeletal muscle mass and function in older adults with sarcopenia. Methodology: Study design: This project will use a pilot 3-arm open-label randomized controlled trial (RCT), designed to evaluate the impact of distinct exercise training regimens on gut microbiome composition in older adults (age ≥ 60 years old) with sarcopenia. Methods: This study will use the recruitment, logistic and material resources from a community exercise program. Those who met our pre-screening criteria will be contacted by a study member, exposing the study's purposes, procedures, risk-discomforts, and benefits. Participants who agree will be invited to an in-person medical screening visit to assess the final inclusion/exclusion criteria and to provide their written informed consent (before enrollment). In this visit, volunteers will be evaluated through clinical examination, medication history, and a handgrip dynamometry test (an objective indicator of sarcopenia) to assess participants eligibility. Those who meet all inclusion/exclusion criteria will be randomly assigned (N= 69; 23/group) to three distinct exercise training programs: i) aerobic exercise (AER) training, ii) resistance exercise (RES), or iii) concurrent training (RES+AER). This project aims to randomize up to n=69 participants (n=23 / group) based on evidence from a recent systematic review with meta-analysis (11). Participants will engage in supervised center-based exercise interventions (12 weeks, 3d/w, 60min/d) consisting of either moderate aerobic training [60-70% HRmax], or resistance exercise [8 exercises/major muscle groups; 6-12 reps; 60-75% 1RM] or a combination of both (RES+AER). Assessments: All participants will be assessed at: i) baseline; ii) end of intervention (14-weeks); and iii) at close-out (26-weeks). Total length of the study is 26-weeks. At each study visit, participants will complete a skeletal muscle strength test, physical performance tests, assessment of body composition and provide a fasted blood, urine and fecal sample. Other important confounding variables will also be recorded including nutritional intake (using a 3-day diary), daily physical activity (using a physical activity tracker- wrist Fitbit), medication and supplementation use and associated comorbidities (assessed through medical and medication history questionnaire). Per the study design, the study team will also evaluate: a) retention and attrition rates; b) adherence to exercise intervention; c) safety; d) intervention effect on dependent outcomes. The success of recruitment and retention rates will be measured by the number of participants recruited, the number of drop-outs and losses to follow-up throughout the trial. Adherence to the exercise intervention will be carefully documented by study staff and will be measured by the number of sessions attended. Safety will be measured by the number and/or seriousness of adverse events attributable to the intervention and monitored and recorded by study staff throughout the trial. Objectives: Primary aim: The primary outcome will be the change in the relative abundance of Faecalibacterium prausnitzii and other SCFA producing bacteria after the intervention (14-weeks). Secondary outcomes include: 1) change of Faecalibacterium prausnitzii relative abundance at close-out (26-weeks); 2) change of relative abundance of Lactobacillus and Bifidobacterium genera after the intervention and at the end of the follow-up. Secondary aim: A set of complementary outcomes will also be assessed to broadly characterize the impact of each exercise intervention, including body composition, skeletal muscle function, functional performance and general gut microbiome composition. This broad set of outcomes will allow a comprehensive evaluation of the impact of these distinct exercise regimens on gut microbiota and on several health outcomes that are crucial for modulating gut microbiome and sarcopenia and may point to other mechanistic links that are currently undetermined. Expected Outcomes: The investigative team hypothesized that combining aerobic and resistance training will have a greater impact on the gut microbiome, specifically in increasing the relative abundance of Faecalibacterium prausnitzii and other SCFA-producing bacterial strains, an increase in skeletal muscle mass and strength, as well as enhanced physical performance measures in the concurrent exercise training group.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 60 years old
* Sex: Men and women
* Medical History: Objective indicators of sarcopenia- Handgrip strength: men < 27 kg and women < 16 kg; 4-m gait speed ≤ 0.8 m/s; Short Physical Performance Battery ≤ 8-point score; Chair stand test > 15 s; Time-up-go ≥ 20 s.
* Physical Inactivity: International Physical Activity Questionnaire (IPAQ)- Portuguese version ≤ 150 minutes/week of moderate physical activity
* Willingness to participate in all study procedures regardless of possible group allocation.

Exclusion Criteria:

* Failure to provide consent.
* Uncontrolled Hypertension: SBP> 180 mmHg or DBP> 110 mmHg.
* History of coronary artery stenosis (>50%).
* Heart Failure: Ejection fraction < 50%.
* History of syncope at exertion.
* History of hypertrophic cardiomyopathy, arrhythmogenic cardiomyopathy, dilated cardiomyopathy or evidence in the previous 6 months of myocarditis or pericarditis.
* Severe valvular heart disease.
* Chronic kidney disease stage ≥ 4,8.
* Chronic Obstructive Pulmonary Disease stage ≥ 3,9.
* Musculoskeletal or neurodegenerative conditions that hinder exercise engagement.
* Current participation in another structured exercise training program.
* Inability to commit to study procedures or the exercise intervention throughout the study period.
* Other condition or concern precluding safe participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Percent change in the relative abundance of Faecalibacterium prausnitzii and other SCFA producing bacteria | 14-weeks
  The primary outcome will be the percent change in the relative abundance of Faecalibacterium prausnitzii and other SCFA producing bacteria after the intervention (14-weeks) using next generation sequencing on faecal samples

SECONDARY OUTCOMES:
Percent change of Faecalibacterium prausnitzii relative abundance at close-out | 26- weeks
  Percent change of Faecalibacterium prausnitzii relative abundance at close-out (26-weeks)using next generation sequencing on faecal samples;
Percent change of relative abundance of Lactobacillus and Bifidobacterium genera after the intervention and at the end of the follow-up | 26- weeks
  Percent change of relative abundance of Lactobacillus and Bifidobacterium genera after the intervention using next generation sequencing on faecal samples

OTHER OUTCOMES:
Body composition | 14- weeks
  Body composition will be assessed by whole-body dual-energy X-ray absorptiometry to measure percent body fat mass, percent lean mass, appendicular lean mass
Skeletal muscle function | 14-weeks
  Dominant lower limb knee extension and flexion muscle strength will be assessed through a isokinetic dynamometer to measure peak torque of extension and flexion total work (J)
Nutritional Intake | 14-weeks
  Participants will be instructed to record all food and beverage intake for three consecutive days using a 3-day food diary prior to the fecal collection day
Physical performance | 14-weeks
  participants will be evaluated using gait speed, the 30-second chair rise, the Short Physical Performance Battery (SPPB) and the 400 meter walk test. To assess gait speed, we will use the 4-meter usual walk test with speed time. The SPPB is a composite test battery that includes assessment of gait speed, a balance test, and a chair stand test. Each test is scored 4 points until a maximum score of 12 points. the 400-meter walk test, participants are asked to complete 20 laps of 20 m, each lap as fast as possible. This test evaluates walking ability and endurance.

CONTACTS AND LOCATIONS:
Overall Officials: Liliana C. Baptista, PhD, Principal Investigator — Faculty of Sport, University of Porto
Locations (1):
- Faculty of Sports, Porto, Portugal

IPD SHARING:
Plan to Share IPD: No
This project contemplates a plan to disseminate knowledge using specific methods and actions, distinct digital platforms and directed to different audiences. The goal is to disseminate the novel findings that may result from this project as soon as possible upon completion and make them publicly available to all that may benefit with it. As soon as the last participant finishes his last assessment visit, the study team members will start to adequately analyze the study data. The study team will prepare abstracts and manuscripts for publication. Preliminary results that may seem adequate for scientific meetings will be prepared in accordance and presented at national or international relevant conferences.

REFERENCES:
- [Derived] Merelim AS, Zacca R, Moreira-Goncalves D, Costa PP, Baptista LC. Distinct exercise modalities on GUT microbiome in sarcopenic older adults: study protocol of a pilot randomized controlled trial. Front Med (Lausanne). 2025 Mar 5;12:1504786. doi: 10.3389/fmed.2025.1504786. eCollection 2025. PMID 40109720